CLINICAL TRIAL: NCT01778504
Title: Diagnosis of Childhood-onset Behavioral Disorders, Neuropsychiatric Disorders and Neurodevelopmental Disorders
Brief Title: Studying Childhood-onset Behavioral, Psychiatric, and Developmental Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130028; 13-M-0028
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-07-08

CONDITIONS: Neuropsychiatric Disorder; Neurological Disorder; Neurodevelopmental Disorder; Sleep
Keywords: Natural History Study; Mental Illness; Autism; Developmental Delay; Genetic Disorder; Natural History
MeSH Terms: conditions — Nervous System Diseases; Neurodevelopmental Disorders; Mental Disorders; Autistic Disorder; Learning Disabilities; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Probands: Children, adolescents, and adults
- Relatives of Probands: 1st, 2nd, and 3rd degree relatives

SUMMARY:
Background:

- Many psychiatric, behavioral, and developmental disorders are genetic. This means that they tend to run in families. Some begin in childhood, while others do not appear until adulthood. Researchers want to look at people of all ages who have these disorders that started in childhood. They will also look at relatives of people with these disorders. This information will allow doctors to learn more about childhood behavioral problems and how they are inherited. It may also help doctors treat those disorders.

Objectives:

- To study the onset and treatment of childhood behavioral, psychiatric, and developmental disorders.

Eligibility:

* Individuals of any age who have a psychiatric, autism spectrum, or developmental disorder, or other behavioral problems.
* Family members of individuals with the above disorders. This group may include parents, grandparents, siblings, aunts/uncles, cousins, and children.

Design:

- Participants will be screened with a medical history and physical exam. They may have a psychiatric history with tests of thinking, judgment, and behavior. Brain imaging scans may be performed to look at brain function.

DETAILED DESCRIPTION:
This is a diagnostic protocol designed to provide opportunities for identifying new clinical syndromes and permitting longitudinal assessments of a variety of childhood behavioral, psychiatric and developmental disorders. Disorders of particular interest are: autism, disorders of social cognition and other neurodevelopmental disorders; childhood psychiatric disorders and particularly those with acute symptom onset; and unique clinical presentations of pediatric behavioral syndromes, such as those associated with genetic disorders or those with a unique family history.

Objectives: The primary objective of this protocol is to evaluate a variety of behavioral, neuropsychiatric, and neurodevelopmental conditions. The protocol will allow OCD investigators to gain additional knowledge about the course of various childhood behavioral syndromes. The information obtained is expected to generate questions to be answered and hypotheses to be tested in future protocols.

Study Population: The number of participants to be enrolled will be set up to 1,000 probands (children, adolescents and adults).

Design: This is a natural history protocol. The cross-sectional portion of this study may include in-depth medical, sleep and neurodevelopmental assessments to evaluate the relationship of biological abnormalities with neuropsychiatric symptomatology. Standard therapeutic interventions may be utilized to evaluate their effects in well-characterized participants with unique clinical presentations. Participants also may be asked to return to NIH for periodic follow-up assessments, in order to facilitate the longitudinal assessment of natural and treated courses of illness as a means of better understanding their progression and pathophysiology.

Outcome Measures: No formal outcomes will be measured; however, the clinical assessments of enrolled participants may be used to evaluate correlates of clinical symptomatology and response to standard therapeutic interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

1. Are aged birth to 99 years
2. Have a diagnosed or undiagnosed neuropsychiatric disorder, neurodevelopmental disability or abnormal behaviors.
3. Have the ability to understand and sign an informed consent on behalf of themselves or their minor children, or have a legal guardian (or designated DPA).
4. Are under the care of a primary physician.

EXCLUSION CRITERIA:

Participants will not be eligible if they:

* Are unwilling or unable to be evaluated and followed as clinically indicated. Examples might include children with severe behavioral problems who refuse physical examination.
* The participant does not have a primary healthcare provider.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 1000 people with psychiatric, behavioral, or developmental disorders will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-12-27 (Actual); Primary Completion 2029-02-20 (Estimated)

PRIMARY OUTCOMES:
clinical assessments | Ongoing
  to evaluate correlates of clinical symptomatology and response to standard therapeutic interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Ashura W Buckley, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Beneke M, Rasmus W. "Clinical Global Impressions" (ECDEU): some critical comments. Pharmacopsychiatry. 1992 Jul;25(4):171-6. doi: 10.1055/s-2007-1014401. PMID 1528956
- [Background] Bodfish JW, Symons FJ, Parker DE, Lewis MH. Varieties of repetitive behavior in autism: comparisons to mental retardation. J Autism Dev Disord. 2000 Jun;30(3):237-43. doi: 10.1023/a:1005596502855. PMID 11055459
- [Background] Constantino JN, Davis SA, Todd RD, Schindler MK, Gross MM, Brophy SL, Metzger LM, Shoushtari CS, Splinter R, Reich W. Validation of a brief quantitative measure of autistic traits: comparison of the social responsiveness scale with the autism diagnostic interview-revised. J Autism Dev Disord. 2003 Aug;33(4):427-33. doi: 10.1023/a:1025014929212. PMID 12959421
- [Derived] Witmer C, Mattingly A, D'Souza P, Thurm A, Hadigan C. Incontinence in Phelan-McDermid Syndrome. J Pediatr Gastroenterol Nutr. 2019 Aug;69(2):e39-e42. doi: 10.1097/MPG.0000000000002342. PMID 30921255
- [Derived] Khan OI, Zhou X, Leon J, Kessler R, Gaughan T, D'Souza P, Gropman A, Cohen N, Rennert O, Buckley A, Inati S, Thurm A. Prospective longitudinal overnight video-EEG evaluation in Phelan-McDermid Syndrome. Epilepsy Behav. 2018 Mar;80:312-320. doi: 10.1016/j.yebeh.2017.11.034. Epub 2018 Feb 3. PMID 29402632
- [Derived] Soorya L, Leon J, Trelles MP, Thurm A. Framework for assessing individuals with rare genetic disorders associated with profound intellectual and multiple disabilities (PIMD): the example of Phelan McDermid Syndrome. Clin Neuropsychol. 2018 Aug-Oct;32(7):1226-1255. doi: 10.1080/13854046.2017.1413211. Epub 2017 Dec 21. PMID 29265961
- [Derived] Gaughan T, Buckley A, Hommer R, Grant P, Williams K, Leckman JF, Swedo SE. Rapid Eye Movement Sleep Abnormalities in Children with Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS). J Clin Sleep Med. 2016 Jul 15;12(7):1027-32. doi: 10.5664/jcsm.5942. PMID 27166296
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-M-0028.html